CLINICAL TRIAL: NCT01852110
Title: A Seamless Phase IIa/IIb, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Trial to Evaluate the Efficacy and Safety of MK-7622 as an Adjunctive Therapy for Symptomatic Treatment in Subjects With Alzheimer's Disease
Brief Title: Efficacy and Safety of MK-7622 as Adjunct Therapy in Participants With Alzheimer's Disease (MK-7622-012)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stage 1 interim analysis of efficacy met the criteria for early trial termination (futility). The trial was terminated at Stage 1; did not proceed to Stage 2.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7622-012; 2013-000937-11 (EudraCT Number); MK-7622-012 (Other: Merck Protocol Number)
Record Dates: First submitted 2013-05-08; First posted 2013-05-13 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- MK-7622 High Dose - 45 mg (Stage 1) (Experimental): Single 45 mg MK-7622 capsule once daily, taken orally. Dose escalated as follows: 15 mg MK-7622 once daily for 1 week; 30 mg MK-7622 once daily for 1 week; and 45 mg MK-7622 once daily for the remainder of treatment.
  Interventions: Drug: MK-7622; Drug: AChEI
- Placebo (Stage 1) (Placebo Comparator): Matching placebo to MK-7622 capsule once daily, taken orally.
  Interventions: Drug: Placebo; Drug: AChEI
- MK-7622 Low Dose - 5 mg (Stage 2) (Experimental): Single 5 mg MK-7622 capsule once daily, taken orally.
  Interventions: Drug: MK-7622; Drug: AChEI
- MK-7622 Mid Dose - 15 mg (Stage 2) (Experimental): Single 15 mg MK-7622 capsule once daily, taken orally.
  Interventions: Drug: MK-7622; Drug: AChEI
- MK-7622 High Dose - 45 mg (Stage 2) (Experimental): Single 45 mg MK-7622 capsule once daily, taken orally. Dose escalated as follows: 15 mg MK-7622 once daily for 1 week; 30 mg MK-7622 once daily for 1 week; and 45 mg MK-7622 once daily for the remainder of treatment.
  Interventions: Drug: MK-7622; Drug: AChEI
- Placebo (Stage 2) (Placebo Comparator): Matching placebo to MK-7622 capsule once daily, taken orally.
  Interventions: Drug: Placebo; Drug: AChEI

INTERVENTIONS:
Drug: MK-7622 — MK-7622 capsule
  Arms: MK-7622 High Dose - 45 mg (Stage 1); MK-7622 High Dose - 45 mg (Stage 2); MK-7622 Low Dose - 5 mg (Stage 2); MK-7622 Mid Dose - 15 mg (Stage 2)
Drug: Placebo — Matching placebo to MK-7622 capsule
  Arms: Placebo (Stage 1); Placebo (Stage 2)
Drug: AChEI — One of the following AChEIs, as prescribed by the participant's primary care physician:
  Donepezil: 10 mg total daily dose, administered orally
  Rivastigmine: 9.5 or 13.3 mg/24 hours, administered by transdermal patch; or 6-12 mg total daily dose administered orally
  Galantamine: 16-24 mg total daily dose, administered orally

SUMMARY:
The purpose of this multicenter trial is to assess the efficacy and safety of MK-7622 compared with placebo as adjunctive therapy to acetylcholinesterase inhibitors (AChEIs) for the symptomatic treatment of participants with mild to moderate Alzheimer's Disease (AD). The trial consists of two stages: Stage 1 and Stage 2. In Stage 1, participants will be randomized to receive either placebo or MK-7622 45 mg once daily. In Stage 2, participants will be randomized to receive either placebo or MK-7622 (dose: 5, 15 or 45 mg once daily). Participants will be enrolled in only one stage; the duration of each stage is approximately 26 weeks. Interim analyses will be performed in both Stage 1 and Stage 2 to determine whether the trial should continue. The primary study hypotheses are the following: Stage 1 - MK-7622 45 mg once daily is superior to placebo with respect to improving cognition in participants with mild to moderate AD as assessed by mean change from baseline in the 11-item Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog11) at Week 12; Stage 2 - At least one of the top two doses of MK-7622 (15 mg once daily, 45 mg once daily) is superior to placebo with respect to improving cognition in participants with mild to moderate AD as assessed by mean change from baseline in ADAS-Cog11 at Week 12.

DETAILED DESCRIPTION:
If the double-blind treatment dose is not tolerated during the first 2 weeks, the participant will be discontinued. After the first 2 weeks, if the dose is not tolerated, the regimen may be modified according to a defined algorithm. Specifically, the participant will begin administration of a reduced dose for up to 2 weeks, followed by a re-challenge at the original dose only if tolerability issues diminish or resolve at the reduced dose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD based on both a) the National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria and b) the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria for AD
* AD is of mild to moderate severity
* Clear history of cognitive and functional decline over at least one year that is either a) documented in medical records or b) documented by history from an informant who knows the participant well
* On a stable and effective daily dose of AChEI (either donepezil, rivastigmine, or galantamine), for at least two months before Screening, and willing to remain on the same dose for the duration of the trial. Effective doses are considered to be: donepezil, 10 mg total daily dose administered orally; rivastigmine, 9.5 or 13.3 mg/24 hours administered by transdermal patch or 6-12 mg total daily dose administered orally; galantamine, 16-24 mg total daily dose administered orally
* Able to read at a 6th grade level or equivalent, and must have a history of academic achievement and/or employment sufficient to exclude mental retardation
* Have a reliable and competent trial partner who must have a close relationship with the subject

Exclusion Criteria:

* History of clinically significant stroke
* Evidence of a neurological disorder other than the disease being studied (i.e., probable AD)
* History of seizures or epilepsy within the last 5 years before Screening
* Evidence of a clinically relevant or unstable psychiatric disorder, excluding major depression in remission
* Is at imminent risk of self-harm or of harm to others
* History of alcoholism or drug dependency/abuse within the last 5 years before Screening
* Does not have a magnetic resonance imaging (MRI) scan obtained within 12 months of Screening and is unwilling or not eligible to undergo an MRI scan at Screening
* History of hepatitis or liver disease that has been active within the six months prior to Screening Visit
* Recent or ongoing, uncontrolled, clinically significant medical condition within 3 months of the Screening Visit (e.g., diabetes, hypertension, thyroid or endocrine disease, congestive heart failure, angina, cardiac or gastrointestinal disease, dialysis, or abnormal renal function) other than the condition being studied such that participation in the trial would pose a significant medical risk to the participant. Controlled co-morbid conditions are not exclusionary if stable within three months of the Screening Visit
* History or current evidence of long QT syndrome, corrected QT (QTc) interval ≥470 milliseconds (for male subjects) or ≥480 milliseconds (for female subjects), or torsades de pointes
* History of malignancy occurring within the five years before Screening, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or localized prostate carcinoma which has been treated with potentially curative therapy with no evidence of recurrence for ≥3 year post-therapy
* Clinically significant vitamin B12 deficiency, or increased thyroid stimulating hormone (TSH) in the six months before Screening
* Major surgery within 3 months of Screening

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-10-22 (Actual); Primary Completion 2016-04-11 (Actual); Study Completion 2016-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Voss T, Li J, Cummings J, Farlow M, Assaid C, Froman S, Leibensperger H, Snow-Adami L, McMahon KB, Egan M, Michelson D. Randomized, controlled, proof-of-concept trial of MK-7622 in Alzheimer's disease. Alzheimers Dement (N Y). 2018 Apr 26;4:173-181. doi: 10.1016/j.trci.2018.03.004. eCollection 2018. PMID 29955661

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Number of Participants Screened: 505 Number of Participants Randomized: 240
Pre-assignment Details: Stage 1 interim analysis met the prespecified futility threshold for the primary efficacy endpoint, satisfying the clinical criteria for early trial termination (futility). As a result, the trial was terminated at Stage 1; did not proceed to Stage 2.
  In stage 1: 1 randomized participant received no study medication (MK-7622 High Dose-45 mg arm).
Period: Overall Study
Arm/Group | MK-7622 High Dose - 45 mg (Stage 1) | Placebo (Stage 1) | MK-7622 Low Dose - 5 mg (Stage 2) | MK-7622 Mid Dose - 15 mg (Stage 2) | MK-7622 High Dose - 45 mg (Stage 2) | Placebo (Stage 2)
Started | 120 | 120 | 0 (Study terminated prior to participant recruitment for Stage 2) | 0 (Study terminated prior to participant recruitment for Stage 2) | 0 (Study terminated prior to participant recruitment for Stage 2) | 0 (Study terminated prior to participant recruitment for Stage 2)
Treated | 119 | 120 | 0 | 0 | 0 | 0
Completed | 70 | 74 | 0 (Study terminated prior to participant recruitment for Stage 2) | 0 (Study terminated prior to participant recruitment for Stage 2) | 0 (Study terminated prior to participant recruitment for Stage 2) | 0 (Study terminated prior to participant recruitment for Stage 2)
Not Completed | 50 | 46 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 12 | 5 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Non-compliance with Study Drug | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 30 | 32 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes only participants in Stage 1 who were both randomized (i.e. started) and treated.
  In stage 1:
  MK-7622 High Dose - 45 mg: of the randomized participants (n=120), all but 1 randomized participant received study treatment (n=119).
  Placebo: Of the randomized participants (n=120), all received study treatment (n=120).
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-7622 High Dose - 45 mg (Stage 1) | Placebo (Stage 1) | Total
Number analyzed (Participants) | 119 | 120 | 239
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.5 (7.1) | 71.7 (8.3) | 72.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 68 | 129
  Male | 58 | 52 | 110
11-item Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog11) Score [Mean (Standard Deviation); unit: Score on a Scale] — ADAS-Cog11 measures cognition by assessing 11 metrics impaired in Alzheimer's Disease (AD): speech; speech comprehension; word finding; word recall; object/finger naming; orientation; obeying commands; ideational praxis; constructional praxis; word recognition; and remembering instruction. For each metric, scores range from 0 (no impairment) to (depending on the metric) either 5 (8 metrics), 8, 10, or 12 (1 metric each); higher scores indicate more severe impairment. Individual scores sum to a total ADAS-Cog11 score (range: 0-70). Higher total scores indicate greater cognitive impairment. Population: Includes only randomized participants receiving ≥1 dose of study medication, having a baseline ADAS-Cog11 assessment.
  Score on a Scale | 21.8 (7.05) | 23.6 (8.73) | 22.7 (7.95)
Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) Score [Mean (Standard Deviation); unit: Score on a Scale] — The ADCS-ADL score measures the performance of activities of daily living, calculated from a 24-question survey. For each of the 24 questions, scores range from 0 (no independence) to (depending on the question) either 2 (1 question), 3 (17 questions), 4 (5 questions), or 5 (1 question), with higher scores indicating greater independence in activity performance. Scores from individual questions are summed into a total ADCS-ADL score, with potential total scores ranging from 0 to 78. Lower scores indicate less independence in activity performance and, as a result, greater AD severity. Population: Includes only randomized participants receiving ≥1 dose of study medication, having a baseline ADCS-ADL assessment.
  Score on a Scale
    number analyzed (Participants) | 119 | 119 | 238
    (all) | 60.7 (11.18) | 59.4 (11.89) | 59.9 (11.72)
Composite Cognition Score-3 Domain (CCS-3D) [Mean (Standard Deviation); unit: z-score] — CCS-3D is composed of individual cognitive tests, grouped into 3 domains: 1) episodic memory; 2) executive function; and 3) attention/processing speed. For each cognitive test, a z-score (Z) is calculated at each time point [Z = (observed value - study population mean at baseline) / study population standard deviation at baseline]. These individual Zs are first combined into domain-specific Zs, and then into a composite Z, (i.e. CCS-3D). Theoretically, 99.9% of CCS-3D will be ± 3; more positive CCS-3D indicate greater cognitive impairment relative to the total study population at baseline. Population: Includes only randomized participants receiving ≥1 dose of study medication, having a baseline CCS-3D assessment.
  z-score
    number analyzed (Participants) | 108 | 110 | 218
    (all) | -0.11 (0.739) | 0.02 (0.816) | -0.039 (0.776)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 11-item Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog11) Score at Week 12 (Stage 1, MK-7622 45 mg Versus Placebo)
Description: Mean change from baseline at week 12 was assessed for ADAS-Cog11 score. ADAS-Cog11 measures cognition by assessing 11 metrics impaired in Alzheimer's Disease (AD): speech; speech comprehension; word finding; word recall; object/finger naming; orientation; obeying commands; ideational praxis; constructional praxis; word recognition; and remembering instruction. For each metric, scores range from 0 (no impairment) to (depending on the metric) either 5 (8 metrics), 8, 10, or 12 (1 metric each); higher scores indicate more severe impairment. Individual scores sum to a total ADAS-Cog11 score, ranging from 0-70. Higher total scores indicate greater cognitive impairment and AD severity. Further, increases in AD severity over time would be reflected by increases in ADAS-Cog11 score.
Time Frame: Baseline and week 12
Population: All randomized participants in Stage 1 receiving ≥1 dose of study medication, having either a baseline or 12-week ADAS-Cog11 assessment.
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | MK-7622 High Dose - 45 mg (Stage 1) | Placebo (Stage 1)
Number analyzed (Participants) | 119 | 120
Score on a Scale | 0.39 (0.440) | 0.21 (0.416)
Statistical Analysis 1: Comparison: MK-7622 High Dose - 45 mg (Stage 1) vs Placebo (Stage 1); Test type: Superiority or Other; p = 0.7623, Constrained Longitudinal Data Analysis; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-1.00 to 1.37]

2. Primary Outcome: Change From Baseline in ADAS-Cog11 Score at Week 12 (Stage 2, MK-7622 45 mg and 15 mg Versus Placebo)
Description: as for outcome 1
Time Frame: Baseline and week 12
Population: Per study protocol, the analysis population was to include only randomized participants in Stage 2 receiving ≥1 dose of placebo, MK-7622 - 15 mg, or MK-7622 - 45 mg, having either a baseline or 12-week ADAS-Cog11 assessment. Study terminated before Stage 2 enrollment; no data were collected for this outcome measure.
Arm/Group | MK-7622 Mid Dose - 15 mg (Stage 2) | MK-7622 High Dose - 45 mg (Stage 2) | Placebo (Stage 2)
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: The number of participants experiencing an adverse event (AE) was assessed. An AE is any unfavorable and unintended medical occurrence, symptom, or disease witnessed in a participant, regardless of whether or not a causal relationship with the study treatment can be demonstrated. Further, any worsening of a preexisting condition that is temporally associated with the use of the study treatment is also considered an AE.
Time Frame: Up to 26 weeks
Population: All participants as treated, consisting of all participants (Stages 1 and 2) who received study medication. Study terminated before Stage 2 enrollment; no data were collected for Stage 2-specific arms.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-7622 High Dose - 45 mg (Stage 1) | Placebo (Stage 1) | MK-7622 Low Dose - 5 mg (Stage 2) | MK-7622 Mid Dose - 15 mg (Stage 2) | MK-7622 High Dose - 45 mg (Stage 2) | Placebo (Stage 2)
Number analyzed (Participants) | 119 | 120 | 0 | 0 | 0 | 0
Participants | 83 | 71 |  |  |  |

4. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: The number of participants discontinuing study drug due to an AE was assessed.
Time Frame: Up to 24 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- MK-7622 Low Dose - 5 mg (Stage 2): Single 5 mg MK-7622 capsule once daily, taken orally, for 24 weeks
Arm/Group | MK-7622 High Dose - 45 mg (Stage 1) | Placebo (Stage 1) | MK-7622 Low Dose - 5 mg (Stage 2) | MK-7622 Mid Dose - 15 mg (Stage 2) | MK-7622 High Dose - 45 mg (Stage 2) | Placebo (Stage 2)
Number analyzed (Participants) | 119 | 120 | 0 | 0 | 0 | 0
Participants | 19 | 7 |  |  |  |

5. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living Inventory (ADCS-ADL) at Week 24 (Combining Stage 1 and 2, MK-7622 45 mg Versus Placebo)
Description: Mean change from baseline at week 24 was assessed for ADCS-ADL score. The ADCS-ADL score measures the performance of activities of daily living, calculated from a 24-question survey. For each of the 24 questions, scores range from 0 (no independence) to (depending on the question) either 2 (1 question), 3 (17 questions), 4 (5 questions), or 5 (1 question), with higher scores indicating greater independence in activity performance. Scores from individual questions are summed into a total ADCS-ADL score, with potential total scores ranging from 0 to 78. Lower scores indicate less independence in activity performance and, as a result, greater AD severity. Further, increases in AD severity over time would be reflected by decreases in ADCS-ADL score.
Time Frame: Baseline and week 24
Population: Per protocol, analysis population was to include all randomized participants (pooled across Stages 1 and 2) receiving ≥1 dose of placebo or MK-7622 - 45 mg, having either a baseline or 24-week ADCS-ADL assessment. As the study was terminated before Stage 2 enrollment, only participants in Stage 1 were analyzed.
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | MK-7622 High Dose - 45 mg (Stage 1) | Placebo (Stage 1)
Number analyzed (Participants) | 119 | 119
Score on a Scale | -2.66 (0.919) | -2.73 (0.853)
Statistical Analysis 1: Comparison: MK-7622 High Dose - 45 mg (Stage 1) vs Placebo (Stage 1); Test type: Superiority or Other; p = 0.9604, Constrained Longitudinal Data Analysis; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-2.42 to 2.54]

6. Secondary Outcome: Change From Baseline in Composite Cognition Score-3 Domain (CCS-3D) at Week 12 (Stage 1, MK-7622 45 mg Versus Placebo)
Description: CCS-3D is composed of individual cognitive tests, grouped into 3 domains: 1) episodic memory; 2) executive function; and 3) attention/processing speed. For each cognitive test, a z-score (Z) is calculated at each time point [Z = (observed value - study population mean at baseline) / study population standard deviation at baseline]. These individual Zs are first combined into domain-specific Zs, and then into a composite Z, (i.e. CCS-3D). Theoretically, 99.9% of CCS-3D will be ± 3; more positive CCS-3D indicate greater cognitive impairment relative to the total study population at baseline. Further, negative changes in CCS-3D over time indicate improved cognition relative to the total study population at baseline.
Time Frame: Baseline and week 12
Population: All randomized participants in Stage 1 receiving ≥1 dose of study medication, having either a baseline or 12-week CCS-3D assessment.
Measure: Mean (Standard Error); unit: z-score
Arm/Group | MK-7622 High Dose - 45 mg (Stage 1) | Placebo (Stage 1)
Number analyzed (Participants) | 108 | 110
z-score | 0.13 (0.043) | 0.03 (0.042)
Statistical Analysis 1: Comparison: MK-7622 High Dose - 45 mg (Stage 1) vs Placebo (Stage 1); Test type: Superiority or Other; p = 0.0829, Constrained Longitudinal Data Analysis; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.01 to 0.22]

7. Secondary Outcome: Change From Baseline in CCS-3D at Week 12 (Stage 2, MK-7622 45 mg and 15 mg Versus Placebo)
Description: as for outcome 6
Time Frame: Baseline and Week 12
Population: Per study protocol, the analysis population was to include only randomized participants in Stage 2 receiving ≥1 dose of placebo, MK-7622 - 15 mg, or MK-7622 - 45 mg, having either a baseline or 12-week CCS-3D assessment. Study terminated before Stage 2 enrollment; no data were collected for this outcome measure.
Arm/Group | MK-7622 Mid Dose - 15 mg (Stage 2) | MK-7622 High Dose - 45 mg (Stage 2) | Placebo (Stage 2)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 26 weeks
Arm/Group | MK-7622 High Dose - 45 mg (Stage 1) | Placebo (Stage 1)
Serious Adverse Events (participants affected / at risk) | 9/119 | 4/120
Other Adverse Events (participants affected / at risk) | 42/119 | 20/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7622 High Dose - 45 mg (Stage 1) (N=119) | Placebo (Stage 1) (N=120)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7622 High Dose - 45 mg (Stage 1) (N=119) | Placebo (Stage 1) (N=120)
Diarrhoea (Gastrointestinal disorders) | 18 (19) | 7 (9)
Urinary tract infection (Infections and infestations) | 6 (7) | 5 (6)
Weight decreased (Investigations) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 11 (12) | 6 (7)
Urinary incontinence (Renal and urinary disorders) | 6 (6) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1)

LIMITATIONS AND CAVEATS:
Stage 1 Interim analysis of efficacy met the clinical criteria for early trial termination (futility). As a result, the trial was terminated at Stage 1 and did not proceed to Stage 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.